CLINICAL TRIAL: NCT06271278
Title: The Effects of Emotional Freedom Technique on Work-Related Stress and Alarm Fatigue in Nurses Working in Surgical Intensive Care Units
Brief Title: The Effect of Emotional Freedom Techniques Application on Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gürkan (Other)
Responsible Party: Sponsor-Investigator, Gürkan, Assistant Professor, Malatya Turgut Ozal University
Organization: Malatya Turgut Ozal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023-17
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Occupational Stress; Alert Fatigue, Health Personnel
Keywords: Surgical intensive care; Alarm Fatigue; Job stress; Emotional Freedom Technique; Surgical nurse
MeSH Terms: conditions — Occupational Stress; Alert Fatigue, Health Personnel

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomised controlled study with experimental and control groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to their group assignment. The subjects will be selected in a randomized order using software. Data collection will be conducted without involvement from research analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Freedom Techniques group (Experimental): The Nurse Introduction Form, Subjective Discomfort Unit, Alarm Fatigue Scale, and Work Stress Scale were administered to the experimental group prior to patient care. The Emotional Freedom Technique was explained, and the nurses were instructed to apply it before and after their shifts for one week. One week later, the Subjective Discomfort Unit, Alarm Fatigue Scale, and Work Stress Scale were applied again.
  Interventions: Behavioral: Emotional Freedom Technique
- Control group (No Intervention): No applications were administered to nurses working in the surgical intensive care unit. In the control group, data was collected before patient care using the Nurse Introduction Form, Subjective Discomfort Unit, Alarm Fatigue Scale, and Work Stress Scale. No interventions were performed. One week later, the Subjective Discomfort Unit, Alarm Fatigue Scale, and Work Stress Scale were applied again.

INTERVENTIONS:
Behavioral: Emotional Freedom Technique — Emotional Freedom Technique (EFT) is a powerful and effective practice that enables individuals to release negative emotions and achieve mental and physical relaxation. EFT is a form of counselling based on acupuncture points, which are areas of low electrical and energy flow in the body. Stimulating these points causes the brain to secrete dopamine. EFT involves stimulating specific points on the body where energy flow is low. This is done by gently tapping on these areas with the fingers, which releases dopamine. The process is painless and can be performed by the individual themselves.
  Arms: Emotional Freedom Techniques group

SUMMARY:
Nurses working in surgical intensive care units face numerous health and safety stressors. The introduction of new health technologies, medical devices (such as bedside monitors, pump and perfuser devices, and mechanical ventilators), and changing health environments have contributed to increased work stress among nurses. This, in turn, has had negative effects on their physical and mental health outcomes. One of the hazards associated with medical devices is alarm fatigue. Noise pollution caused by bells, beeps, and horns in intensive care units can lead to alarm fatigue, defined as desensitisation to monitor alarms. Nurses are particularly susceptible to this due to their constant exposure to these sounds, which can also cause stress. Occupational stress is a recognised issue in this demanding field, characterised by disproportionate workloads and negative effects on performance.Work-related stress can lead to a loss of compassion towards patients and an increase in malpractice, negatively affecting the quality of care. Thus, this study aimed to investigate the impact of applying emotional freedom techniques on work-related stress and alarm fatigue experienced by nurses working in surgical intensive care units.

DETAILED DESCRIPTION:
Surgical intensive care units have high mortality and mobility rates and require 24-hour monitoring. Intensive care environments are stressful for working individuals, particularly nurses, due to health and safety concerns. In recent years, new health technologies and medical devices, as well as changing health environments, have increased work stress among nurses, leading to negative physical and mental health outcomes. The use of medical device alarms, including bedside monitors, pump devices, perfuser devices, patient heating-cooling devices, mechanical ventilators, computers, and nutrition devices, has increased over time. These alarms are used to monitor changes in the vital signs of patients and ensure continuity of care. However, alarm fatigue is a significant problem caused by medical devices. Noise pollution is a common issue in intensive care units due to the various sounds emitted by medical devices. Health professionals may experience alarm fatigue, which is defined as desensitisation to monitor alarms. Dealing with alarm fatigue requires objective and comprehensible solutions. Inappropriate techniques such as disabling alarms, delayed response, setting them between unsafe parameters, and turning down the volume so low that they cannot be heard, are cognitive stressors. The continuous exposure to these alarm sounds, coupled with the nature of nurses' work, can also cause stress. Occupational stress is a demanding profession that can have negative effects on performance. Therefore, it is important to address occupational stress in the nursing profession. It is quite common among nurses and can jeopardise both their quality of life and patient safety. Work-related stress can lead to a loss of compassion towards patients and an increase in malpractice, negatively affecting the quality of care. Thus, this study aimed to investigate the impact of applying emotional freedom techniques on work-related stress and alarm fatigue experienced by nurses working in surgical intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Working as a nurse in one of the surgical intensive care units
* Volunteering to participate in the study

Exclusion Criteria:

* Working in a unit other than surgical intensive care units
* Not volunteering to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Disturbance Scale | 0-7 days tracking
  The discomfort scale used in energy therapies allows individuals to evaluate their own discomfort on a scale of 0 to 10, where 0 indicates no discomfort and 10 indicates unbearable discomfort.
Alarm Fatigue Scale | 0-7 days tracking
  The scale consists of 13 items and produces a score between 0 and 36. A higher score indicates an increase in alarm fatigue.
The General Work Stress Scale | 0-7 days tracking
  The General Work Stress Scale is a 9-item scale that produces scores ranging from 9 to 45. High scores indicate high job stress, while low scores indicate low job stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University Turgut OzaL Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No